CLINICAL TRIAL: NCT00042432
Title: A Study of an Investigational Medication for Secondary Hyperparathyroidism in Chronic Renal Insufficiency Patients
Brief Title: Study for Secondary Hyperparathyroidism in Chronic Renal Insufficiency Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20010239
Record Dates: First submitted 2002-07-29; First posted 2002-08-01 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Secondary Hyperparathyroidism; Chronic Renal Insufficiency
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- cinacalcet (AMG 073) (Experimental)
  Interventions: Drug: cinacalcet (AMG 073)
- Placebo (Placebo Comparator)
  Interventions: Drug: cinacalcet (AMG 073)

INTERVENTIONS:
Drug: cinacalcet (AMG 073) — Initially receive 1 tablet of study medication (cinacalcet or placebo) once daily. Possible sequential dose titrations are 30, 60, 90, 120, 180mg cinacalcet or placebo) daily. The titration phase was 12 weeks and the efficacy assessment phase was 6 weeks.

SUMMARY:
This study will assess an investigational medication for patients with chronic renal insufficiency (pre-dialysis) who have secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have chronic renal insufficiency (pre-dialysis)
* Have below normal creatinine clearance
* Have elevated parathyroid hormone levels

Exclusion Criteria:

* Pregnant or nursing
* Heart attack in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2002-06; Primary Completion 2003-03 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Charytan C, Coburn JW, Chonchol M, Herman J, Lien YH, Liu W, Klassen PS, McCary LC, Pichette V. Cinacalcet hydrochloride is an effective treatment for secondary hyperparathyroidism in patients with CKD not receiving dialysis. Am J Kidney Dis. 2005 Jul;46(1):58-67. doi: 10.1053/j.ajkd.2005.04.013. PMID 15983958
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 28 June 2002 through 14 November 2002
Groups:
- Cinacalcet (AMG 073): Cinacalcet administered orally once daily with dose titrated starting at 30 mg
- Placebo: Placebo administered orally once daily
Period: Overall Study
Arm/Group | Cinacalcet (AMG 073) | Placebo
Started | 27 | 27
Completed | 18 | 20
Not Completed | 9 | 7
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Death | 0 | 2
Not completed — Ineligibility determined | 1 | 0
Not completed — Initiation of maintenance dialysis | 1 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cinacalcet (AMG 073) | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (15.5) | 61.9 (15.2) | 61.2 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 16 | 22 | 38
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 18 | 13 | 31
  Black | 6 | 10 | 16
  Other | 3 | 4 | 7
Glomerular Filtration Rate (GFR) Stratification Factor [Number; unit: Participants]
  GFR ≥ 15 and < 25 ml/min/1.73 m^2 | 20 | 19 | 39
  GFR ≥ 25 and ≤ 50 ml/min/1.73 m^2 | 7 | 8 | 15
Intact Parathyroid Hormone (iPTH) [Mean (Standard Deviation); unit: pg/mL] | 243.3 (139.5) | 236.1 (189.5) | 239.7 (164.9)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Mean iPTH of ≥ 30% During the Efficacy Assessment Phase
Description: Reduction in mean intact parathyroid hormone (iPTH) of ≥ 30% within the participant during the efficacy assessment phase
Time Frame: Efficacy assessment phase (weeks 12-18)
Population: All randomized participants, using Last Value Carried Forward (LVCF) imputation
Measure: Number; unit: Participants
Arm/Group | Cinacalcet (AMG 073) | Placebo
Number analyzed (Participants) | 27 | 27
Participants | 15 | 5
Statistical Analysis 1: Comparison: Cinacalcet (AMG 073) vs Placebo; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; Adjusted for baseline glomenular filtration rate (GFR) strata; Odds Ratio (OR) = 5.67, 95% CI [1.60 to 20.06] — Logit estimates

2. Secondary Outcome: Percentage Change From Baseline in Mean iPTH During the Efficacy Assessment Phase
Description: Percentage change from baseline in mean intact parathyroid hormone (iPTH) during the efficacy assessment phase
Time Frame: Baseline, efficacy assessment phase (weeks 12-18)
Population: All randomized participants, using Last Value Carried Forward (LVCF) imputation
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Cinacalcet (AMG 073) | Placebo
Number analyzed (Participants) | 27 | 27
Percent change | -31.5 (6.70) | 5.8 (6.97)
Statistical Analysis 1: Comparison: Cinacalcet (AMG 073) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Adusted for baseline glomerular filtration rate (GFR) strata

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 6/27 | 3/27
Other Adverse Events (participants affected / at risk) | 20/27 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Cinacalcet (N=27)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Cinacalcet (N=27)
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 2 | 9
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 2 | 1
Chills (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 3 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 4 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.